CLINICAL TRIAL: NCT01226823
Title: Intrahepatic Cholestasis Of Pregnancy: Clinical Impact Of Ursodeoxycholic Acid Treatment
Brief Title: Ursodeoxycholic Acid And Cholestasis Of Pregnancy
Acronym: CERTO
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Modified insurance requests by a new law released after its approval.
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Francesco Azzaroli, Assistant Professor, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CERTO
Record Dates: First submitted 2010-10-19; First posted 2010-10-22 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Intrahepatic Cholestasis of Pregnancy
Keywords: cholestasis; pregnancy; ursodeoxycholic acid; ICP
MeSH Terms: conditions — Intrahepatic Cholestasis of Pregnancy; Cholestasis | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): obstetrical monitoring plus placebo
  Interventions: Drug: Placebo
- Ursodeoxycholic acid (Experimental): obstetrical monitoring plus active drug
  Interventions: Drug: Ursodeoxycholic Acid

INTERVENTIONS:
Drug: Ursodeoxycholic Acid — 300 mg capsules 20 mg/kg body weight/day divided in three administrations per day from enrolment until delivery
  Arms: Ursodeoxycholic acid
Drug: Placebo — 300 mg capsules 20 mg/kg body weight/day divided in three administrations per day from enrolment until delivery
  Arms: Placebo

SUMMARY:
The study is a multicenter randomized double blind placebo controlled trial. The study will be conducted on pregnant women with a diagnosis of intrahepatic cholestasis of pregnancy (ICP) in third level hospitals (that are also Academic Hospitals).

Pregnant women at the time of ICP diagnosis will be randomized in two groups:

Group 1 - will receive placebo and obstetrical monitoring until delivery Group 2 - will receive UDCA at the dose of 20 mg/Kg/day and obstetrical monitoring until delivery.

The hypotheses are that UDCA treatment will be superior to placebo and effective in:

reducing the rate of prematurity; improving maternal biochemical parameters and symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant state (after week 20 of gestation)
* Total Serum BA elevation (>10 micromol/l)
* Transaminases elevation (ALT>40 UI/L and AST>37 UI/L)
* Occurrence of pruritus
* Informed consent signed

Exclusion Criteria:

* Infectious diseases (HBV, HDV, HCV related liver disease, EBV, CMV, HIV infection)
* Dermatologic diseases
* Metabolic diseases (including alcohol abuse)
* Other causes of cholestasis (i.e. PBC; PSC)
* Autoimmune liver disease
* Obstructive biliary diseases
* Drug related pathologies
* Known or suspected hyper-sensibility to the drug or the pharmacological class under study
* Serious clinical conditions that, according to the judgment of the investigator, contraindicate the participation to the study (heart, kidney and liver disease)
* Use of cholestyramine
* Patients not able or not willing to follow the procedures of the protocol
* Patients not signing the informed consent
* Onset of ICP during of after the 36th week of pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-11; Primary Completion 2013-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with preterm delivery (before week 37) | at the time of delivery

SECONDARY OUTCOMES:
Pruritus on the Visual Analogue Scale | from enrollment until delivery
Transaminases | from enrolment until delivery
Bile Acids | from enrolment until delivery
Fetal movement count | from enrolment until delivery
  mother evaluation
Number of pregnancies with cardiotocography suggestive of fetal stress | from enrolment until delivery
APGAR index | 1 and 5 minutes after birth
Number of pregnancies with Green stained amniotic fluid | at delivery
  obstetrician evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Mazzella, Professor, Study Director — University of Bologna; Francesco Azzaroli, Professor, Principal Investigator — University of Bologna
Locations (7):
- Italy (7):
  - Divisione di Gastroenterologia, IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - Dept. of Surgical and Gastroenterological Sciences, University of Padova, Padua, Italy
  - UOC Ostetricia e Ginecologia, Ospedale Maggiore, Bologna
  - S.Orsola-Malpighi Hospital, Bologna
  - Gastroenterology and Liver Clinic, Azienda Ospedaliero-Universitaria, University of Modena and Reggio Emilia, Modena
  - Gastroenterology Unit, Policlinic of Palermo, Palermo
  - Internal Medicine Department, Gemelli Hospital, Catholic University of Sacred Heart, Rome

REFERENCES:
- [Derived] Walker KF, Chappell LC, Hague WM, Middleton P, Thornton JG. Pharmacological interventions for treating intrahepatic cholestasis of pregnancy. Cochrane Database Syst Rev. 2020 Jul 27;7(7):CD000493. doi: 10.1002/14651858.CD000493.pub3. PMID 32716060